CLINICAL TRIAL: NCT01095796
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Elvitegravir/Emtricitabine/Tenofovir Disoproxil Fumarate/GS-9350 Versus Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Brief Title: Study to Evaluate the Safety and Efficacy of Stribild Versus Atripla in Human Immunodeficiency Virus, Type 1 (HIV-1) Infected, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-236-0102
Record Dates: First submitted 2010-03-17; First posted 2010-03-30 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: HIV; HIV Infections
Keywords: Treatment Naive; HIV 1 Infected
MeSH Terms: conditions — HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stribild (Experimental): Stribild plus placebo to match Atripla
  Interventions: Drug: Stribild; Drug: Atripla Placebo
- Atripla (Active Comparator): Atripla plus placebo to match Stribild
  Interventions: Drug: Atripla; Drug: Stribild Placebo

INTERVENTIONS:
Drug: Stribild — Stribild (EVG 150 mg/COBI 150 mg/FTC 200 mg/TDF 300 mg) STR administered orally once daily
  Arms: Stribild
Drug: Atripla — Atripla (EFV 600 mg/FTC 200 mg/TDF 300 mg) tablet administered orally once daily prior to bedtime
  Arms: Atripla
Drug: Stribild Placebo — Placebo to match Stribild STR administered orally once daily
  Arms: Atripla
Drug: Atripla Placebo — Placebo to match Atripla tablet administered orally once daily prior to bedtime
  Arms: Stribild

SUMMARY:
To evaluate the safety and efficacy of Stribild®, a single tablet regimen (STR) containing fixed doses of elvitegravir (EVG)/cobicistat (COBI [GS-9350])/emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) versus efavirenz (EFV)/FTC/TDF (Atripla®) in HIV-1 infected, antiretroviral treatment-naive adults. Stribild offers an alternative STR for patients who are not candidates for non-nucleoside reverse transcriptor-based STRs.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* Plasma HIV-1 RNA levels ≥ 5,000 copies/mL
* No prior use of any approved or investigational antiretroviral drug for any length of time
* Screening genotype report must show sensitivity to FTC, TDF, and EFV
* Normal electrocardiogram (ECG)
* Adequate renal function (estimated glomerular filtration rate ≥ 70 mL/min according to the Cockcroft Gault formula)
* Hepatic transaminases (aspartate aminotransferase (AST) and alanine aminotransferase (ALT)) ≤ 5 x the upper limit of the normal range (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Serum amylase ≤ 5 x ULN
* Males and females of childbearing potential must agree to utilize highly effective contraception methods from screening throughout the duration of study treatment and for 12 weeks following the last dose of study drug
* Age ≥ 18 years
* Life expectancy ≥ 1 year

Exclusion Criteria:

* A new acquired immunodeficiency syndrome (AIDS)-defining condition diagnosed within the 30 days prior to screening
* Receiving drug treatment for hepatitis C, or anticipated to receive treatment for hepatitis C
* Subjects experiencing decompensated cirrhosis
* Females who are breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Implanted defibrillator or pacemaker
* Current alcohol or substance use judged by the Investigator to potentially interfere with subject study compliance
* History of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, noninvasive cutaneous squamous carcinoma
* Active, serious infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Medications contraindicated for use with EVG, COBI, FTC, EFV, or TDF; or subjects with any known allergies to the excipients of Stribild or Atripla tablets
* Participation in any other clinical trial without prior approval
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rhee, MD, Study Director — Gilead Sciences
Locations (102):
- United States (97):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - Health for Life Clinic PLLC, Little Rock, Arkansas
  - AHF Research Center, Beverly Hills, California
  - Kaiser Permanente Hospital, Hayward, California
  - Living Hope Clinical Foundation, Long Beach, California
  - Kaiser Permanente, Los Angeles, California
  - Los Angeles Gay and Lesbian Center DBA Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - UCLA Center for Clinical Aids Research and Education, Los Angeles, California
  - Peter J. Ruane, MD, Inc., Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Anthony Mills, MD, Inc., Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - Alameda County Medical Center, Oakland, California
  - East Bay AIDS Center, Oakland, California
  - Stanford University, Palo Alto, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - San Francisco General Hospital, University of California, San Francisco, San Francisco, California
  - Metropolis Medical, San Francisco, California
  - Kaiser Permanente Medical Center, Clinical Trials Unit, San Francisco, California
  - Apex Research, LLC, Denver, Colorado
  - Yale University HIV Clinical Trials Program, New Haven, Connecticut
  - The Stamford Hospital, Stamford, Connecticut
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Broward Health/Comprehensive Care Center, Fort Lauderdale, Florida
  - Gary J. Richmond, MD, PA, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - The Kinder Medical Group, Miami, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Idocf/ Valuhealthmd, Llc, Orlando, Florida
  - University of South Florida HIV Clinical Research Unit / Hillsborough County Health Department, Tampa, Florida
  - Infectious Disease Research Institute Inc., Tampa, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Atlanta ID Group, PC, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - Leahi Hospital, Honolulu, Hawaii
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Community Research Initiative, Boston, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Baystate Infectious Diseases Clinical Research, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Central West Clinical Research, St Louis, Missouri
  - Southampton Healthcare, St Louis, Missouri
  - ID Care, Hillsborough, New Jersey
  - Saint Michaels Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Garden State Infectious Diseases Associates, PA, Voorhees Township, New Jersey
  - SouthWest CARE Center, Sante Fe, New Mexico
  - Upstate ID Association, Albany, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Hospital Queens, Flushing, New York
  - North Shore University Hospital, Manhasset, New York
  - Greiger Clinic, Mount Vernon, New York
  - Beth Israel Medical Center, New York, New York
  - Chelsea Village Medical, PC, New York, New York
  - Ricky K. Hsu, MD, PC, New York, New York
  - The Aaron Diamond AIDS Research Center, New York, New York
  - Montefiore Medical Center - AIDS Center, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - Clinical and Translational Research Center, Chapel Hill, North Carolina
  - Carolinas Medical Center-Myers Park, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - University of South Carolina, Columbia, South Carolina
  - Southwest Infectious Disease Clinical Research, Inc., Dallas, Texas
  - Peabody Health Center, Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Valley AIDS Council, Harlingen, Texas
  - Therapeutic Concepts, Houston, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - Research Access Network, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education, Infectious Diseases (CARE-ID), Annandale, Virginia
  - Peter Shalit, MD, Seattle, Washington
  - Rockwood Pulmonary and Critical Care, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Puerto Rico (5):
  - Instituto de Investigacion Clentifica del Sur, Ponce
  - Clinical Research Puerto Rico, San Juan
  - HOPE Clinical Research, San Juan
  - VA Caribbean Healthcare System, San Juan
  - University of Puerto Rico, School of Medicine, Proyecto ACTU, San Juan

REFERENCES:
- [Result] Sax PE, DeJesus E, Mills A, Zolopa A, Cohen C, Wohl D, Gallant JE, Liu HC, Zhong L, Yale K, White K, Kearney BP, Szwarcberg J, Quirk E, Cheng AK; GS-US-236-0102 study team. Co-formulated elvitegravir, cobicistat, emtricitabine, and tenofovir versus co-formulated efavirenz, emtricitabine, and tenofovir for initial treatment of HIV-1 infection: a randomised, double-blind, phase 3 trial, analysis of results after 48 weeks. Lancet. 2012 Jun 30;379(9835):2439-2448. doi: 10.1016/S0140-6736(12)60917-9. PMID 22748591
- [Result] Zolopa A, Sax PE, DeJesus E, Mills A, Cohen C, Wohl D, Gallant JE, Liu HC, Plummer A, White KL, Cheng AK, Rhee MS, Szwarcberg J; GS-US-236-0102 Study Team. A randomized double-blind comparison of coformulated elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate versus efavirenz/emtricitabine/tenofovir disoproxil fumarate for initial treatment of HIV-1 infection: analysis of week 96 results. J Acquir Immune Defic Syndr. 2013 May 1;63(1):96-100. doi: 10.1097/QAI.0b013e318289545c. PMID 23392460
- [Result] Wohl DA, Cohen C, Gallant JE, Mills A, Sax PE, Dejesus E, Zolopa A, Liu HC, Plummer A, White KL, Cheng AK, Rhee MS, Szwarcberg J; GS-US-236-0102 Study Team. A randomized, double-blind comparison of single-tablet regimen elvitegravir/cobicistat/emtricitabine/tenofovir DF versus single-tablet regimen efavirenz/emtricitabine/tenofovir DF for initial treatment of HIV-1 infection: analysis of week 144 results. J Acquir Immune Defic Syndr. 2014 Mar 1;65(3):e118-20. doi: 10.1097/QAI.0000000000000057. No abstract available. PMID 24256630

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at sites in the United States and Puerto Rico. The first participant was screened on 16 March 2010. The last study visit occurred on 02 September 2014.
Pre-assignment Details: 917 participants were screened.
Groups:
- Stribild: Stribild® (elvitegravir (EVG) 150 mg/cobicistat (COBI) 150 mg/emtricitabine (FTC) 200 mg/tenofovir disoproxil fumarate (TDF) 300 mg) single-tablet regimen (STR) once daily plus placebo to match Atripla once daily prior to bedtime
- Atripla: Atripla® (efavirenz (EFV) 600 mg/FTC 200 mg/TDF 300 mg) tablet once daily prior to bedtime plus placebo to match Stribild once daily
Period: Overall Study
Arm/Group | Stribild | Atripla
Started | 353 | 354
Completed | 58 | 65
Not Completed | 295 | 289
Not completed — Randomized but Not Treated | 5 | 2
Not completed — Adverse Event | 9 | 19
Not completed — Death | 3 | 2
Not completed — Pregnancy | 2 | 0
Not completed — Lack of Efficacy | 5 | 3
Not completed — Investigator's Discretion | 7 | 2
Not completed — Withdrew Consent | 16 | 22
Not completed — Lost to Follow-up | 27 | 29
Not completed — Participant Noncompliance | 5 | 10
Not completed — Protocol Violation | 1 | 0
Not completed — Participant Transferred to Another Study | 215 | 200

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least one dose of study medication.
Groups:
- Stribild: Stribild (EVG 150 mg/COBI 150 mg/FTC 200 mg/TDF 300 mg) STR once daily plus placebo to match Atripla once daily prior to bedtime
- Atripla: Atripla (EFV 600 mg/FTC 200 mg/TDF 300 mg) tablet once daily prior to bedtime plus placebo to match Stribild once daily
- Total: Total of all reporting groups
Arm/Group | Stribild | Atripla | Total
Number analyzed (Participants) | 348 | 352 | 700
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (10.4) | 38 (10.6) | 38 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 36 | 77
  Male | 307 | 316 | 623
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 6 | 10 | 16
  Black or African Heritage | 106 | 91 | 197
  Native Hawaiian or Pacific Islander | 4 | 1 | 5
  White | 214 | 227 | 441
  Other | 16 | 19 | 35
Region of Enrollment [Number; unit: participants]
  United States | 348 | 352 | 700
HIV Disease Status [Number; unit: participants]
  Asymptomatic | 290 | 295 | 585
  Symptomatic HIV Infections | 30 | 33 | 63
  AIDS | 28 | 24 | 52
Hepatitis B Virus (HBV) Infection Status [Number; unit: participants]
  Negative | 343 | 343 | 686
  Positive | 5 | 9 | 14
Hepatitis C Virus (HCV) Infection Status [Number; unit: participants]
  Negative | 331 | 337 | 668
  Positive | 17 | 15 | 32
HIV-1 RNA Category (copies/mL) [Number; unit: participants]
  ≤ 100,000 | 230 | 236 | 466
  > 100,000 | 118 | 116 | 234
CD4 Cell Count (/µL) [Number; unit: participants]
  ≤ 50 | 7 | 6 | 13
  51 to ≤ 200 | 36 | 45 | 81
  201 to ≤ 350 | 112 | 96 | 208
  351 to ≤ 500 | 113 | 136 | 249
  > 500 | 80 | 69 | 149

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Virologic Success Using the Food and Drug Administration (FDA)-Defined Snapshot Analysis as Determined by the Achievement of HIV-1 Ribonucleic Acid (RNA) < 50 Copies/mL at Week 48
Time Frame: Week 48
Population: Intent-to-treat (ITT) Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 348 | 352
percentage of participants | 87.6 | 84.1
Statistical Analysis 1: Comparison: Stribild vs Atripla; The null hypothesis was that the percentage of participants achieving HIV-1 RNA < 50 copies/mL (as defined by the snapshot analysis algorithm) at Week 48 in the Stribild group is at least 12% worse than the response rate in the Atripla group; the alternative hypothesis was that the response rate in the Stribild group is less than 12% worse than that in the Atripla Group; Test type: Non-Inferiority or Equivalence — A total of 700 HIV-1 infected participants, randomized in a 1:1 ratio to 2 groups would achieve at least 95% power to establish noninferiority in Week 48 response (HIV-1 RNA < 50 copies/mL per the FDA-defined snapshot analysis) rate difference between the 2 groups. For sample size and power computation, it was assumed that both treatment groups have a response rate of 0.795, a noninferiority margin of 0.12, and that the significance level of the test is at a one-sided, 0.025 level; Difference in response rates = 3.6, 95.2% CI 2-sided [-1.6 to 8.8] — To preserve the overall alpha level: 0.05, accounting for 2 interim analyses for Independent Data Monitoring Committee meetings, the 95.2% CI was computed using normal approximation stratified by baseline HIV-1 RNA (≤ 100,000 or > 100,000 copies/mL)

2. Secondary Outcome: The Percentage of Participants With Virologic Success Using the FDA-Defined Snapshot Analysis as Determined by the Achievement of HIV-1 RNA < 50 Copies/mL at Week 96
Time Frame: Week 96
Population: ITT Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 348 | 352
percentage of participants | 84.2 | 81.5

3. Secondary Outcome: The Percentage of Participants With Virologic Success Using the FDA-Defined Snapshot Analysis as Determined by the Achievement of HIV-1 RNA < 50 Copies/mL at Week 144
Time Frame: Week 144
Population: ITT Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 348 | 352
percentage of participants | 80.2 | 75.3

4. Secondary Outcome: The Percentage of Participants With Virologic Success Using the FDA-Defined Snapshot Analysis as Determined by the Achievement of HIV-1 RNA < 50 Copies/mL at Week 192
Time Frame: Week 192
Population: Week 192 Modified Intent-to-treat (MITT) Analysis Set: Participants in the ITT analysis set, excluding those who either 1) transferred to other Gilead-sponsored studies after completing their Week 144 Visit and before the lower limit of the Week 192 analysis window, or 2) prematurely discontinued study drug prior to the Week 144 Visit.
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 71 | 73
percentage of participants | 76.1 | 78.1

5. Secondary Outcome: The Percentage of Participants Achieving and Maintaining Confirmed HIV-1 RNA < 50 Copies/mL at Week 48 Using the FDA-defined Time to Loss of Virologic Response (TLOVR) Algorithm
Time Frame: Week 48
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 348 | 352
percentage of participants | 85.9 | 83.2

6. Secondary Outcome: The Change From Baseline in Cluster Determinant 4 (CD4) Cell Count at Weeks 48, 96, 144, and 192
Description: Change = value of the relevant time point minus the baseline value
Time Frame: Baseline; Weeks 48, 96, 144, and 192
Population: ITT Analysis Set. The missing = excluded (M = E) method was used in which all participants with missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 348 | 352
cells/µL
  Change at Wk 48 (Stribild, n=325; Atripla, n=315) | 239 (167.2) | 206 (153.4)
  Change at Wk 96 (Stribild, n=307; Atripla, n=302) | 295 (213.3) | 273 (189.7)
  Change at Wk 144 (Stribild, n=294; Atripla, n=283) | 321 (227.0) | 300 (202.3)
  Change at Wk 192 (Stribild, n=62; Atripla, n=69) | 360 (285.9) | 328 (227.6)

7. Secondary Outcome: The Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Time Frame: Week 48
Population: ITT Analysis Set. The missing = failure (M = F) method was used in which all missing data were considered as failure (HIV-1 RNA ≥ 50 copies/mL).
Measure: Number; unit: percentage of participants
Arm/Group | Stribild | Atripla
Number analyzed (Participants) | 348 | 352
percentage of participants | 88.8 | 85.5

ADVERSE EVENTS:
Time Frame: Up to 218 weeks plus 30 days
Description: Safety Analysis Set: participants were randomized and received at least one dose of study drug.
Arm/Group | Stribild | Atripla
Serious Adverse Events (participants affected / at risk) | 69/348 | 50/352
Other Adverse Events (participants affected / at risk) | 313/348 | 326/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (N=348) | Atripla (N=352)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 | 1
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Intracardiac mass (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal mass (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 4 | 3
Bronchitis (Infections and infestations) | 1 | 3
Bronchitis bacterial (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 6 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Giardiasis (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0
Muscle abscess (Infections and infestations) | 1 | 0
Neurosyphilis (Infections and infestations) | 1 | 2
Ovarian abscess (Infections and infestations) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 9 | 2
Pneumonia legionella (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Secondary syphilis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 3 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anorectal human papilloma virus infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Immune reconstitution inflammatory syndrome associated Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Convulsion (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Alcoholism (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 1
Completed suicide (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 2 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Drug dependence (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Testicular mass (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Alcohol use (Social circumstances) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stribild (N=348) | Atripla (N=352)
Lymphadenopathy (Blood and lymphatic system disorders) | 16 | 18
Abdominal pain (Gastrointestinal disorders) | 24 | 18
Constipation (Gastrointestinal disorders) | 22 | 14
Diarrhoea (Gastrointestinal disorders) | 93 | 91
Dyspepsia (Gastrointestinal disorders) | 19 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19 | 14
Haemorrhoids (Gastrointestinal disorders) | 23 | 13
Nausea (Gastrointestinal disorders) | 80 | 59
Vomiting (Gastrointestinal disorders) | 28 | 23
Fatigue (General disorders) | 53 | 61
Pyrexia (General disorders) | 21 | 23
Bronchitis (Infections and infestations) | 41 | 37
Chlamydial infection (Infections and infestations) | 23 | 13
Folliculitis (Infections and infestations) | 17 | 18
Gonorrhoea (Infections and infestations) | 22 | 9
Herpes zoster (Infections and infestations) | 19 | 9
Influenza (Infections and infestations) | 15 | 19
Nasopharyngitis (Infections and infestations) | 38 | 34
Pharyngitis (Infections and infestations) | 16 | 22
Sinusitis (Infections and infestations) | 41 | 46
Syphilis (Infections and infestations) | 34 | 33
Upper respiratory tract infection (Infections and infestations) | 92 | 78
Decreased appetite (Metabolism and nutrition disorders) | 18 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 24
Anorectal human papilloma virus infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 13
Dizziness (Nervous system disorders) | 29 | 94
Headache (Nervous system disorders) | 62 | 45
Somnolence (Nervous system disorders) | 7 | 28
Abnormal dreams (Psychiatric disorders) | 56 | 101
Anxiety (Psychiatric disorders) | 30 | 33
Depression (Psychiatric disorders) | 56 | 59
Insomnia (Psychiatric disorders) | 47 | 63
Erectile dysfunction (Reproductive system and breast disorders) | 13 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 26
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 32
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 22 | 14
Dermatitis (Skin and subcutaneous tissue disorders) | 16 | 20
Rash (Skin and subcutaneous tissue disorders) | 35 | 53
Hypertension (Vascular disorders) | 21 | 22

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years